CLINICAL TRIAL: NCT01658787
Title: 'GREAT' Global Registry for Endovascular Aortic Treatment - Outcomes Evaluation
Brief Title: Global Registry for Endovascular Aortic Treatment (GREAT)
Acronym: GREAT
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: GRT 10-11
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Multiple Pathologies
Keywords: Aorta
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endovascular aortic repair: Patients treated with Gore Endovascular Aortic Products.
  Interventions: Device: Endovascular aortic repair

INTERVENTIONS:
Device: Endovascular aortic repair — Treatment with Gore Endovascular Aortic Products.

SUMMARY:
Prospective, observational Registry to obtain data on device performance and clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective observational cohort Registry designed to obtain data on device performance and clinical outcomes of patients treated with Gore Endovascular Aortic products.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age required by state regulations
* Indication for aortic endovascular stent graft repair
* Signed informed consent

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive series of patients who undergo treatment with Gore endovascular aortic products.
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To collect "real world" data on the incidence of serious device events. | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ross Milner, MD, FACS, Principal Investigator — The University of Chicago Medicine & Biological Sciences; Dennis Gable, MD, Principal Investigator — Baylor Research Institute; Pierre Galvagni Silveira, MD, PhD, Principal Investigator — Coris Medicina Avançada; Steven R Dubenec, MD, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia; Santi Trimarchi, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (6):
- United States (2):
  - The University of Chicago Medicine & Biological Sciences, Chicago, Illinois
  - Baylor Research Institute, Plano, Texas
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- Coris Medicina Avançada, Florianópolis, Brazil
- Italy (2):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Policlinico San Donato, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grassi V, Trimarchi S, Weaver F, de Beaufort HWL, Azzizzadeh A, Upchurch GR Jr, Piffaretti G, Lomazzi C; GREAT participants. Endovascular repair of descending thoracic aortic aneurysms-a mid-term report from the Global Registry for Endovascular Aortic Treatment (GREAT). Eur J Cardiothorac Surg. 2022 Jan 24;61(2):357-364. doi: 10.1093/ejcts/ezab366. PMID 34392333
- [Derived] Baxter RD, Hansen SK, Gable CE, DiMaio JM, Shutze WP, Gable DR; GREAT Investigators. Outcomes of Open Versus Percutaneous Access for Patients Enrolled in the GREAT Registry. Ann Vasc Surg. 2021 Jan;70:370-377. doi: 10.1016/j.avsg.2020.06.033. Epub 2020 Jun 27. PMID 32603847
- [Derived] Piffaretti G, Grassi V, Lomazzi C, Brinkman WT, Navarro TP, Jenkins MP, Trimarchi S; GREAT participants. Thoracic endovascular stent graft repair for ascending aortic diseases. J Vasc Surg. 2019 Nov;70(5):1384-1389.e1. doi: 10.1016/j.jvs.2019.01.075. Epub 2019 May 21. PMID 31126763
- [Derived] Shutze W, Suominen V, Jordan W, Cao P, Oweida S, Milner R. The incidence and effect of noncylindrical neck morphology on outcomes after endovascular aortic aneurysm repair in the Global Registry for Endovascular Aortic Treatment. J Vasc Surg. 2018 Dec;68(6):1714-1724. doi: 10.1016/j.jvs.2018.03.394. Epub 2018 May 24. PMID 29803683
- [Derived] Briggs C, Babrowski T, Skelly C, Milner R. Anatomic and clinical characterization of the narrow distal aorta and implications after endovascular aneurysm repair. J Vasc Surg. 2018 Oct;68(4):1030-1038.e1. doi: 10.1016/j.jvs.2017.12.073. Epub 2018 May 22. PMID 29802041